CLINICAL TRIAL: NCT05512156
Title: Toothbrushing Program in Saudi Arabia "TOPS"- A Cluster Randomized Controlled Trial in Kindergartens, Riyadh
Brief Title: Toothbrushing Program in Saudi Arabia "TOPS"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Budur Almutairi, Principal Investigator, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 200263-41
Record Dates: First submitted 2022-08-10; First posted 2022-08-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Dental Caries in Children
Keywords: caries; children; prevention; toothbrushing; kindergartens
MeSH Terms: interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): All children in the intervention arm of the study will be receiving daily supervised toothbrushing in kindergartens for two years. All children are exposed to background water fluoridation.
  Interventions: Other: Supervised Toothbrushing
- Control Group (No Intervention): All children in the control arm of the study will be receiving TAU which is awareness sessions in the school about importance of the daily brushing, healthy diet and demonstrating how to brush correctly and efficiently. All children are exposed to background water fluoridation.

INTERVENTIONS:
Other: Supervised Toothbrushing — * Recruitment, consent, and Questionnaires (Behaviors, Quality of Live, Cost Analysis) distribution.
  * Inclusion & Exclusion Criteria Applied
  * Baseline Dental examination
  * Toothbrushes & Toothpastes Home and school use packs delivery-Colgate (six pack per child a year- child soft toothbrush with a1450ppm fluoridated toothpaste))
  * Supervised teachers training
  * Three months intervals monitoring visits
  * "12months" Follow up and Questionnaires (Behaviours) distribution
  * Endpoint dental Examination and Questionnaires (Behaviours, Quality of Live, Cost Analysis) distribution
  Other Names: toothbrushing
  Arms: Intervention Group

SUMMARY:
Project summary

Introduction: Dental caries is a major oral health problem worldwide and is a particular public health challenge in Saudi Arabia. Dental caries cause pain, infection, and negatively impact quality of life. As part of population oral health improvement efforts in Saudi Arabia, this project aims to evaluate the effectiveness of a supervised toothbrushing programme in kindergartens.

Aim: The aim of this project is to conduct a trial to assess the effectiveness of a supervised toothbrushing programme in kindergartens in Riyadh, Saudi Arabia .

Methods: A cluster randomized controlled trial study will be undertaken in which the effectiveness of the daily supervised toothbrushing programme intervention running for two academic years will be randomly allocated to a sample of kindergartens in Riyadh and compared against treatment as usual which will be an annual oral health awareness visit in the control group of kindergartens over and above community water fluoridation. Effectiveness will be measured and delivered in terms of preventing dental caries in children when compared with children in the treatment as usual control group receiving the same level of community water fluoridation, but not the toothbrushing program intervention.

All children in all kindergartens (both intervention and control groups) will have a dental examination (via trained and calibrated dental teams recording dental caries levels via dmft index) at baseline before intervention commences and at two academic years. In addition, questionnaires on behaviours and quality of life. In addition, process monitoring, and cost analysis surveys will be distributed.

Research Questions:

* Can such a supervised toothbrushing programme in kindergartens be effective at reducing the development of dental caries by 6 years of age?
* Can a supervised toothbrushing programme in kindergartens in Saudi Arabia be established and implemented?

DETAILED DESCRIPTION:
Background Studies confirmed caries and socio-economic factors association. Caries prevalence in children was related to parental factors, such as parents' socio-economic status, behaviors, and their attitudes to oral health. Several studies examined the prevalence of dental caries and associated social risk factors among preschool children in Riyadh, Saudi Arabia. Al-Meedani and Al-Dlaigan in 2016, found that among the total of 388 children examined in Riyadh, 69% had dental caries. There was no statistically significant difference between boys and girls in caries prevalence. There was a significant association between caries prevalence and parental educational level. Children of mothers with postgraduate degrees had higher caries prevalence of 57% while children of mothers with bachelor's degrees and high school level or below had caries prevalence of 66% and 78% respectively. The children of non-working parents had higher caries prevalence compared to those with working parents. The children from larger family size had higher caries prevalence as compared to those from smaller family size.

Another study by Wyne (2008) reported an overall caries prevalence of 74.8% among preschool children who had a mean age of 4.7 years in Riyadh. Similarly, Al-Malik et al (2003) found that 73% of two- to five-year-old children in Saudi Arabia were diagnosed with caries4. Another cross-sectional study by AlMarshad et al 2021, included Saudi preschoolers aged 36-71 months where a total of 383 children were examined. Early childhood caries (ECC) prevalence was 72.6%. Children from schools in northern Riyadh and those of fathers in professional jobs were less likely to have ECC. Children with a nocturnal feeding history and poor oral hygiene were more likely to have ECC.

Oral health improvement programms in education settings such as kindergartens and schools are particularly important because they have shown to be effective and can have the potential of a wide reach across the population during the crucial early years of childhood. Some studies have found that a programme of supervised daily toothbrushing in school can be effective in caries reduction particularly in high-risk populations, it can reduce caries increment in a population experiencing high levels of dental disease. In addition, school-based supervised toothbrushing programme can improve oral hygiene including decreasing levels of plaque, gingival bleeding, and gingivitis. There have been fewer randomized controlled trials of supervised toothbrushing programme particularly in areas with high caries or where other oral health improvement program or initiatives are in place such as water fluoridation.

In a trial including 2228 two to four year-old children attending kindergartens in two counties in northern Hesse, German were randomly allocated to participate in daily tooth brushing with 500 ppm fluoride toothpaste, which was supervised by specially trained dental nurses. The caries increment of the test group was 24% lower than the increment of the control group, and high increment values were observed in the control group twice as often as in the test group. Another trial in England recruited a total of 517 children (mean age 5.63 years) which children in the intervention group brushed once a day at school. For children in the intervention group, the overall caries increment (2.60) was significantly less than for children in the non-intervention group (2.92). In Kaunas city of Lithuania a sample of 411 three years old children were selected to participate in the prevention programme. For test group, supervised toothbrushing was prescribed, and for the control group, children did not undergo any of the procedures. The prevalence of dental caries varied between 39.7% and 90.8%, the reduction in test group was 45.4%. In another clinical trial in Tayside, that was to determine the reduction in two-year caries increment that can be achieved by daily supervised toothbrushing on schooldays, combined with recommended daily home use, compared to a control group involving no intervention. A sample of 534 children, mean age 5.3, in schools in deprived areas were recruited and significant reductions of 32% at D (1) and 56% at D (3) were found. In a study in Jordan, has a similar cultural and community background to Saudi Arabia, caries status of children in the supervised daily tooth brushing group over four years was better than that of the control group. The difference was statistically significant with estimates of relative risk values also showed that children in the control group are 3.1 and 6.4 times at higher risk of having dental caries than those in the study group for age group 12 and six respectively .

Although, there were no enough studies undertaken in background of water fluoridation or in the Saudi population, many international good studies for long follow-up periods had recommended to apply the supervised toothbrushing programme especially in communities with a high prevalence of caries, such as the Saudi community.

Study rationale - hypothesis In kindergartens schools in Saudi Arabia - the main setting for this trial - despite the extremely high levels of dental caries among young children attending, there has been no oral health improvement program established to date.

This trial will assess whether a supervised toothbrushing program can be established and implemented and what the barriers and facilitators to roll out would be. It also aims to deliver direct benefits to the trial population by reducing caries prevalence. The null hypothesis is therefore that the caries levels of children in the supervised toothbrushing arm of the trial after two academic years of the intervention will be no different to that of the children in the control arm. The intervention is also taking place in areas where there has been community water fluoridation since 2007.

Study objectives The objective of this study is to compare the effectiveness of supervised toothbrushing with treatment as usual in preventing any further dental decay from developing.

Methods/Design Basic Design: Cluster randomized of tooth-brushing in kindergartens in Riyadh KSA Group 1 - Toothbrushing. Group 2 - Leaflet. Definition of endpoints and covariates The main outcome measurement will be the number of teeth with obvious decay experience into the dentine for a participating child. This will be measured at both the baseline visit and after two years of follow up. The difference from two years minus the baseline measure will then be calculated. Any negative differences will be set to zero. Negative differences can happen either due to tooth trauma or due to variations in the inspection data (which is to be expected due to the nature of tooth charting, and this is especially possible when different dentists/therapists inspect the same child). The primary endpoint will be 'worsening of decay', namely an increase in the number of decayed teeth of one or more. This variable can be coded as a binary variable with categories of Yes and No. The secondary endpoint will be the increase in the number of teeth affected. The study will recruit from both public and private kindergartens. A priori subgroups of region, school type and the sex of the child will be considered. A further subgroup of existing decay at baseline (Yes/No) will be considered.

Study population One hundred fifty-three children will be recruited into each of the two arms of the study. They will be identified in 20 kindergartens public and private schools in the Riyadh city, North and East areas. The sample is four years old attending participating kindergartens schools. Children approval to participate will be assessed by consent forms that will be send to parents and schools prior to study entry.

Inclusion criteria

* Receipt of a signed informed consent form from a parent or legal guardian.
* Children in the second year of kindergarten school (known as KG2).
* Children with or without pre-existing dental caries.

Exclusion criteria

_ Child is unwell on the same day of dental inspection.

Identification of participants and consent Once the head teacher has given permission, a consent form will be given or sent to the parents or guardians of every KG2 child. Informed consent will be obtained directly by members of the study team at their child' s kindergarten or advance consent arranged by the headteacher. On the day of the dental inspection any child showing distress or verbal, or non-verbal signs of extreme reluctance will be excluded from the study if the dentists feel that continuing with the inspection would cause the child further distress.

Study schedule Up to three visits are involved for children who are retained throughout the study. The first will be to complete the baseline dental inspection and baseline questionnaires distribution. The second visit is after one year of intervention for follow up, toothbrushing packs and behavioral questionnaires distribution. The final visit is to undertake an endpoint dental inspection to reinspect the child in year three of their kindergarten school and endpoint questionnaires distribution. Neither children nor parents are required to make special visits to a clinic or other study base.

Visit 1: Examination /0-month intervention visit(s) At this visit study staff will confirm eligibility before the baseline dental examination is carried out by a study dental practitioner (e.g., signed consent form is in place, and the child has no obvious temporary infections or injuries which would lead to exclusion on the day). Completion of dental examination data and then packages of toothbrushes will be distributed, and supervised toothbrushing will be explained to both teachers and children follow to Childsmile guidelines.

Visit 2: One academic year (+/- 3 months) Questionnaires and toothbrushing packs distribution.

Visit 3: Two academic years (+/- 3 months) Endpoint Questionaries' distribution and end-of-study dental examination visit.

This visit will be conducted when participating children are in KG3, and and approximately five to six years old. The final dental examination will be carried out, regardless of whether the sequence of the supervised toothbrushing had been interrupted or discontinued for any reason.

Study outcome measures The main outcome measurement will be the number of teeth with obvious decay experienced into dentine for a participating child. This will be measured at both the baseline visit and after two academic years of follow-up. The difference from two academic years minus the baseline measure will then be calculated. Any negative differences will be set to zero. Negative differences can happen either due to tooth trauma or due to variations in the inspection data. This is to be expected due to the nature of tooth charting, and this is especially possible when different dentists/therapists inspect the same child.

The primary endpoint will be 'worsening of decay', namely an increase in the number of decayed, missing, or filled teeth of one or more. This variable can be coded as a binary variable with categories of Yes and No. The secondary endpoint will be the increase in the number of teeth affected.

Sample size The sample size calculation is based on the primary endpoint of decay worsening. This calculation has used a power of 80% and an alpha level of 5%. As this is a cluster randomized trial the usual sample size is slightly inflated by the design effect (DE) of DE = 1 + (N - 1) *ICC. N is the average class size, which assumed to be 15 children being successfully inspected. Partly based on pilot data and partly based on the traditionally weak intra-class correlations (ICC) in public health that have been assumed to be 0.001, which produces a DE of 1.019. To detect a difference of 15% worsening in the toothbrushing group versus 30% in the leaflet group,122 children in each group with evaluable endpoints will be required, providing a total sample size of 244 children. Note that to contribute an evaluable endpoint a child will need valid dental inspections at both the baseline and the end of the study. However, in practice not all the children will complete the study. If a loss to follow-up rate of 20% assumed, inflation of the number of children are required to be randomized to153 in each group, and 306 children in total. This corresponds to approximately 20 schools.

In summary:

* randomize 153+153 = 306, from 10+10 schools,
* the sample size requires 122+122 = 244 evaluable endpoints.

Withdrawal of subjects Parents who withdraw their child will be asked, if appropriate, to agree to their having the end-of-study dental examination, to make best use of the information that has been collected on that child. Children who leave a trial kindergarten school during the study, but remain in the local area, and go on to attend a local school will receive an endpoint dental inspection. The parents/guardians of these children will be informed of the inspection. Any adverse reactions to the fluoride (e.g., mucositis, allergic reaction etc.), whether noted by dental staff or reported by parents or school, will be entered into the Case Report Form by the study team. All recorded adverse reactions will be reviewed and if any immediate adverse reaction is suspected, the toothpaste can be easily removed by toothbrushing, rinsing and spitting. In the event of a child having to leave the study due to withdrawn consent, or moving home and so on, the head teacher at the school will inform the study team. If the parent agrees, arrangements will be made to complete the end-of-study dental inspection to maintain that child in the study database (End of Study Form completed).

Statistics and data analysis The primary endpoint of Worsening Decay will be tabulated and analyzed by odds-ratios, with the attendant 95% confidence interval and p-value. This will also be carried out for the three subgroups separately. Additionally, interaction tests will look at any possible synergy or antagonism of the treatment effect with the three subgroups (separately). Logistic regression models will be used for these analyses. The numeric value of the number of excess teeth with obvious decay (i.e., the secondary endpoint) will also be analyzed. All statistical tests will be carried out at the traditional 5% significance level, using the software package SAS version 9.4. There are no issues with multiple testing as the primary endpoint and analysis are clearly defined, with the other analyses being of an exploratory nature.

Questionnaires In addition to clinical data, information on how a child's general and oral health affect their quality of life will be collected using a Child Health Utility 9D questionaries' which will be distributed at three points in the trial: at baseline,12 months and endpoint .Also, parents/guardians of participants will be asked to complete behavioural questionnaire on how is the health of child teeth, how they take care of them and the child diet, in baseline,12months and endpoint intervals(APPENDIX 8) and, a questionnaire on health and dental care services resource use (APPENDIX 9) designed to elicit information on uptake of health and dental care services and medication use by the child within the past 12 months will also be at each of the baseline and endpoint rounds. The questionnaire packs will be distributed to the families via the kindergarten. Follow-up procedures parental questionnaire survey, several well-established techniques to enhance response rates will be used.

These are:

* the cover page for the questionnaire pack sent at baseline.
* parents who had previously provided a mobile telephone number will receive a text reminder if they have not returned the questionnaires within one week.
* at the end of the second week a second copy of the questionnaire pack will be mailed to any non-responders directly to their home address or distributed via the child's kindergarten.
* at the end of the third week the non-responder parent will be contacted by telephone to remind them to complete the questionnaires.

In addition, information on school health policies about School Health Services, school physical environment, School Health Services, health education, school policies and Resources will be collected through headteachers surveys(APPENDIX 10).

Intervention Costs Staff travel costs that are related to staff delivering the interventions will be collected. Members of staff will be asked to fill in a "staff travel cost" form each time they visit a kindergarten. A full economic evaluation of the study will be carried out and will be reported separately following the UK's National Institute for Health and Care Excellence (NICE) public health economic evaluation guidelines, [NICE, 2012]. Health outcomes will be expressed over the two academic years follow-up period using the Child Health Utility 9 Dimensions questionnaire to obtain utility scores.

Intervention Group

* Recruitment, consent, and Questionnaires (Behaviours, Quality of Live, Cost Analysis) distribution.
* Inclusion & Exclusion Criteria Applied
* Baseline Dental examination
* Toothbrushes & Toothpastes packs delivery (six pack per child a year- child soft toothbrush with a1450ppm fluoridated toothpaste))
* Supervised teachers training
* Three months intervals monitoring visits
* "12months" Follow up and Questionnaires (Behaviours) distribution
* Endpoint dental Examination and Questionnaires (Behaviours, Quality of Live, Cost Analysis) distribution

Dry Toothbrushing

* The supervisor should wash their hands with soap and warm water, and thoroughly dry them, before and after the toothbrushing session to prevent cross-infection.
* The child (under supervision) is responsible for collecting the toothbrush from the storage system. Adaptations should be considered if a child has additional support needs.
* Toothpaste is dispensed following the appropriate methods
* Toothpaste provided by the program, containing 1,450 ppm (parts per million) fluoride, is used.
* A pea-sized amount for children three years and over.
* Where toothpaste is shared, a supervisor dispenses it onto a clean surface such as a plate or paper towel.
* There is sufficient spacing between the quantities of dispensed toothpaste to allow collection without cross-contamination.
* Toothpaste must only be dispensed at the time the child is ready to brush.
* Supervisors should cover any cuts, abrasions or breaks in their skin with a waterproof dressing.
* Children may be seated or standing while toothbrushing takes place.
* After toothbrushing is completed, children should spit excess toothpaste into either a disposable tissue, disposable paper towel or disposable cup.
* Tissues/paper towels or cups must be disposed of immediately after use in a bin.
* Toothbrushes can either be returned to the storage system by each child. The system is then taken to an identified sink area by the supervisor, who is responsible for rinsing each toothbrush individually under cold running water or rinsed at a designated sink area where each child is responsible for rinsing their own toothbrush under cold running water. The supervisor or the child can be responsible for the control of the running tap.
* After rinsing of the toothbrushes is complete, the child or the supervisor is responsible for shaking off excess water into the sink. Toothbrushes should not come into contact with the sink.
* Each child (under supervision) is responsible for returning their own toothbrush to the storage system to air dry. Adaptations should be considered if a child has additional support needs. Lids should be replaced at this stage if there is sufficient air circulation.
* Paper towels should be used to mop up all visible drips on the storage system.
* Children should be supervised. It can be done by lines or sitting on their chairs to be better controlled.
* Supervisors are responsible for cleaning sinks with disinfectant after toothbrushing is completed.

Control Group:

All children in the control arm of the study will be receiving TAU which is awareness sessions in the school about importance of the daily brushing, healthy diet and demonstrating how to brush correctly and efficiently. All children are exposed to background water fluoridation.

Study Monitoring Study Monitoring Visits will be conducted by the Saudi Ministry of Health (MOH) dental staff team every three months with toothbrushing packet distribution. A monitoring sheet will be used by the monitor and the supervised teacher. A single named person at each treatment site, responsible for overseeing the intervention, will be asked on each quarterly visit whether children have the opportunity to brush their teeth every day, and if not to explain when/why this may not be possible. They will then be asked to give the main challenges to daily brushing (barriers) and to say what helps.

Process evaluation

Research team will conduct an integrated process evaluation of the trial, which will allow us to:

* Describe the implementation of the intervention and data collection in schools, including barriers and facilitators to efficiency and effectiveness
* Collate experiences of those involved, including staff and parents
* Make recommendations for full roll-out of the program in Saudi Arabia, should the trial be successful
* Make recommendations for the carrying out of trials in early years settings, and for complex community-based trials in general

Monitoring visits Process visits to treatment sites will take place quarterly (every three months) throughout the trial. These will be carried out by the MOH dental team staff and will coincide with delivery/ distribution of trial materials (toothbrushing packs) for efficiency of cost.

A single named person at each treatment site, responsible for overseeing the intervention, will be asked on each quarterly visit whether children have the opportunity to brush their teeth every day, and if no to explain when/why this may not be possible. They will then be asked to give main challenges to daily brushing (barriers) and to say what helps (facilitators; see Appendix 11, part B, the dedicated pro-forma to assess uptake/fidelity of the intervention).

Context surveys As well as quarterly monitoring visits, a dedicated survey of school health policies and practices will be carried out. This survey will be administered to Head Teachers (or other suitable education leads) at both treatment and control schools. This covers any ongoing contextual activity that could affect the children's oral health such as hygiene provision, nutritional services and policies, health education and resources etc.

The process evaluation is guided by a simple logic model for the trial which sets out intended resource use, key activities and intended short and longer-term outcomes.

Training and calibration course The training and calibration course for the Detailed dmft survey of KG2 children in Riyadh will be organized and held by Dental Health Department-Health at MOH in Sep,2022. The training and calibration protocol and materials follows the Scottish National Dental Inspection program resources NDIP. Mandatory training and calibration will run three inspection teams (three dentists and three dental assistants). Training involves sessions on inspection procedures, tooth codes and diagnostic criteria based on the British Association for the Study of Community Dentistry (BASCD) Trainers' Pack5. Clinical training sessions will then undertake on schoolchildren and will be followed by the calibration sessions on a further group of KG2 children. Calibration sessions involve each inspection team examining the same children. The number of children on each course range from 11 to 12. Analyses will be then undertaken by the Community Oral Health research group, University of Glasgow Dental School. Inter-examiner agreement will then be assessed using the percentage agreement and Kappa statistic assessed at the tooth level on dmft components.

Ethical considerations This study was approved ethically by the King Fahad Medical City institutional review board in the Saudi Ministry of Health (22-083E/March 2022). Study participants will only be allowed to enter the study once either a parent or legal guardian has provided written informed consent. The Chief Investigator will be responsible for updating the Ethics Committee on any latest information that is related to the study. The data analysis for this study had been approved ethically by the University of Glasgow Medicine, Veterinary, and Life Sciences Research Ethical Committee (200220194/March 2023).

Informed consent Written informed consent will be obtained from a parent or legal guardian, as applicable, of each trial participant. When a study team member present at the kindergarten will explain the exact nature of the study, answer any questions, and address any concerns. Trial participants will be informed that they are free to withdraw their consent from the study at any time.

Dissemination of findings Study team members will collaborate on producing papers to be submitted to peer-reviewed journals and abstracts of proposed presentations at national and international conferences and symposia.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of a signed informed consent form from a parent or legal guardian.
* Children in the second year of kindergarten school (known as KG2).
* Children with or without pre-existing dental caries.

Exclusion Criteria:

-Child is unwell on the same day of dental inspection.

Ages: 42 Months to 66 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 588 (Actual)
Dates: Start 2022-09-18 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Dental caries using dmft score dental inspection | 2 years
  worsening of decay will be tabulated and analysed by odds-ratios, with the attendant 95% confidence interval and p-value.

SECONDARY OUTCOMES:
The numeric value of the number of excess teeth with obvious decay | 2 years
  (i.e., the secondary endpoint) will also be analysed. All statistical tests will be carried out at the traditional 5% significance level, using the software package SAS version 9.4.

CONTACTS AND LOCATIONS:
Locations (1):
- Saudi Ministry of Health, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Data sharing Is any of the data suitable for sharing? Trial data will be available after publication of primary results. How will the data be shared? File transfer protocol Who should be able to access and use the shared data? Collaboration by application

REFERENCES:
- [Background] Borges HC, Garbin CA, Saliba O, Saliba NA, Moimaz SA. Socio-behavioral factors influence prevalence and severity of dental caries in children with primary dentition. Braz Oral Res. 2012 Nov-Dec;26(6):564-70. doi: 10.1590/s1806-83242012000600013. PMID 23184168
- [Background] Al-Meedani LA, Al-Dlaigan YH. Prevalence of dental caries and associated social risk factors among preschool children in Riyadh, Saudi Arabia. Pak J Med Sci. 2016 Mar-Apr;32(2):452-6. doi: 10.12669/pjms.322.9439. PMID 27182260
- [Background] Wyne AH. Caries prevalence, severity, and pattern in preschool children. J Contemp Dent Pract. 2008 Mar 1;9(3):24-31. PMID 18335116
- [Background] Al-Malik MI, Holt RD, Bedi R. Prevalence and patterns of caries, rampant caries, and oral health in two- to five-year-old children in Saudi Arabia. J Dent Child (Chic). 2003 Sep-Dec;70(3):235-42. PMID 14998208
- [Background] AlMarshad LK, Wyne AH, AlJobair AM. Early childhood caries prevalence and associated risk factors among Saudi preschool children in Riyadh. Saudi Dent J. 2021 Dec;33(8):1084-1090. doi: 10.1016/j.sdentj.2021.04.003. Epub 2021 Apr 21. PMID 34938053
- [Background] Clark E, Foster Page LA, Larkins K, Leon de la Barra S, Murray Thomson W. Caries-preventive efficacy of a supervised school toothbrushing programme in Northland, New Zealand. Community Dent Health. 2019 Feb 25;36(1):9-16. doi: 10.1922/CDH_4337Clark08. PMID 30667188
- [Background] Borges-Yanez SA, Castrejon-Perez RC, Camacho MEI. Effect of a School-Based Supervised Tooth Brushing Program In Mexico City: A Cluster Randomized Intervention. J Clin Pediatr Dent. 2017;41(3):204-213. doi: 10.17796/1053-4628-41.3.204. PMID 28422600
- [Background] Pieper K, Winter J, Krutisch M, Volkner-Stetefeld P, Jablonski-Momeni A. Prevention in kindergartens with 500 ppm fluoride toothpaste-a randomized clinical trial. Clin Oral Investig. 2016 Jul;20(6):1159-64. doi: 10.1007/s00784-015-1604-3. Epub 2015 Sep 23. PMID 26395351
- [Background] Jackson RJ, Newman HN, Smart GJ, Stokes E, Hogan JI, Brown C, Seres J. The effects of a supervised toothbrushing programme on the caries increment of primary school children, initially aged 5-6 years. Caries Res. 2005 Mar-Apr;39(2):108-15. doi: 10.1159/000083155. PMID 15741722
- [Background] Andruskeviciene V, Milciuviene S, Bendoraitiene E, Saldunaite K, Vasiliauskiene I, Slabsinskiene E, Narbutaite J. Oral health status and effectiveness of caries prevention programme in kindergartens in Kaunas city (Lithuania). Oral Health Prev Dent. 2008;6(4):343-8. PMID 19178101
- [Background] Curnow MM, Pine CM, Burnside G, Nicholson JA, Chesters RK, Huntington E. A randomised controlled trial of the efficacy of supervised toothbrushing in high-caries-risk children. Caries Res. 2002 Jul-Aug;36(4):294-300. doi: 10.1159/000063925. PMID 12218280
- [Background] Al-Jundi SH, Hammad M, Alwaeli H. The efficacy of a school-based caries preventive program: a 4-year study. Int J Dent Hyg. 2006 Feb;4(1):30-4. doi: 10.1111/j.1601-5037.2006.00156.x. PMID 16451437
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Derived] Almutairi B, Conway D, Ross A, Hattan M, Almogren F, McMahon AD. Toothbrushing programme in Saudi Arabia 'TOPS': a study protocol for a cluster randomised controlled trial in kindergartens, Riyadh. BMJ Open. 2024 Aug 3;14(8):e083504. doi: 10.1136/bmjopen-2023-083504. PMID 39097315